CLINICAL TRIAL: NCT01627808
Title: Study on Fluid Optimization in Liver Surgery Trough Vigileo/FloTac System Associated to Traditional Monitoring.
Brief Title: Fluid Optimization in Liver Surgery
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Germano De Cosmo, Phd, Catholic University of the Sacred Heart
Other Study IDs: 656/11
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Cancer of Liver
Keywords: intraoperative monitoring; fluid management
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to analyze hemodynamic changes, in patients undergoing liver resection, through the Vigileo/FloTrac system.

DETAILED DESCRIPTION:
To reduce bleeding, hepatectomies are performed with low central pressure (CVP) combined with extrahepatic control flow.

This management can lead hemodynamic instability and reduction in oxygen delivery so an advanced monitoring should be used.

This study analyzes hemodynamic changes, in patients undergoing liver resection, through the Vigileo/FloTrac system.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III

Exclusion Criteria:

* Cirrhosis
* systolic ventricular contractility or diastolic relaxation alterations
* ischemic or valvular diseases
* absence of sinusal rhythm
* impaired renal function

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study were enrolled patients scheduled for elective major hepatic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Stroke volume variation | at time of surgery
  Evaluation of changes in Stroke Volume Variation from Vigileo/FloTrac system during liver resection.

SECONDARY OUTCOMES:
Stroke volume variation | at the end of surgery
  Evaluation of changes in Stroke Volume Variation at the end of liver resection, during fluid optimization.

CONTACTS AND LOCATIONS:
Overall Officials: Germano De Cosmo, PhD, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred heart, Rome, Italy

REFERENCES:
- [Background] Stephenson KR, Steinberg SM, Hughes KS, Vetto JT, Sugarbaker PH, Chang AE. Perioperative blood transfusions are associated with decreased time to recurrence and decreased survival after resection of colorectal liver metastases. Ann Surg. 1988 Dec;208(6):679-87. doi: 10.1097/00000658-198812000-00002. PMID 3196088
- [Background] Torzilli G, Makuuchi M, Inoue K. The vascular control in liver resection: revisitation of a controversial issue. Hepatogastroenterology. 2002 Jan-Feb;49(43):28-31. PMID 11941976
- [Background] Smyrniotis V, Kostopanagiotou G, Theodoraki K, Tsantoulas D, Contis JC. The role of central venous pressure and type of vascular control in blood loss during major liver resections. Am J Surg. 2004 Mar;187(3):398-402. doi: 10.1016/j.amjsurg.2003.12.001. PMID 15006570
- [Background] Chouker A, Schachtner T, Schauer R, Dugas M, Lohe F, Martignoni A, Pollwein B, Niklas M, Rau HG, Jauch KW, Peter K, Thiel M. Effects of Pringle manoeuvre and ischaemic preconditioning on haemodynamic stability in patients undergoing elective hepatectomy: a randomized trial. Br J Anaesth. 2004 Aug;93(2):204-11. doi: 10.1093/bja/aeh195. Epub 2004 Jun 11. PMID 15194628
- [Background] Bein B, Worthmann F, Tonner PH, Paris A, Steinfath M, Hedderich J, Scholz J. Comparison of esophageal Doppler, pulse contour analysis, and real-time pulmonary artery thermodilution for the continuous measurement of cardiac output. J Cardiothorac Vasc Anesth. 2004 Apr;18(2):185-9. doi: 10.1053/j.jvca.2004.01.025. PMID 15073709
- [Background] Hickey R. How good is arterial pulse contour (LiDCO) and the esophageal Doppler monitor (HemoSonic) in measuring left ventricular stroke volume during venous occlusion? Crit Care Med. 2008 Nov;36(11):3103-4. doi: 10.1097/CCM.0b013e31818b927a. No abstract available. PMID 18941314
- [Background] Mayer J, Boldt J, Mengistu AM, Rohm KD, Suttner S. Goal-directed intraoperative therapy based on autocalibrated arterial pressure waveform analysis reduces hospital stay in high-risk surgical patients: a randomized, controlled trial. Crit Care. 2010;14(1):R18. doi: 10.1186/cc8875. Epub 2010 Feb 15. PMID 20156348
- [Background] Marquez J, McCurry K, Severyn DA, Pinsky MR. Ability of pulse power, esophageal Doppler, and arterial pulse pressure to estimate rapid changes in stroke volume in humans. Crit Care Med. 2008 Nov;36(11):3001-7. doi: 10.1097/CCM.0b013e31818b31f0. PMID 18824912